CLINICAL TRIAL: NCT03741478
Title: Effect of Antipsychotics on Central Insulin Action in Relation to Glucose Metabolism and Cognition in Healthy Volunteers
Brief Title: Intranasal Insulin and Olanzapine Study in Healthy Volunteers
Acronym: INI/OLA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Margaret Hahn, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 075/2017
Record Dates: First submitted 2018-11-03; First posted 2018-11-15 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Olanzapine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study will follow a single-blind, crossover design wherein each participant will participate in all of the possible treatment combinations including:
  Cognitive Arm:
  1. Intranasal placebo and placebo
  2. Intranasal placebo and olanzapine
  3. Intranasal insulin and placebo
  4. Intranasal insulin and olanzapine
  Metabolic Arm:
  1. Intranasal placebo and placebo
  2. Intranasal insulin and placebo
  3. Intranasal insulin and olanzapine
Who Masked: Participant, Investigator
Masking Description: Participants will be masked to:
  1. Knowing whether they were assigned to the olanzapine or placebo conditions
  2. Knowing whether they were assigned to the intranasal insulin or intranasal placebo conditions.
  Investigators will only be masked to the randomization of placebo or olanzapine for the participants, but will know whether the participant receives intranasal insulin or intranasal placebo. In the Cognitive Arm, a separate staff member who is unaware of drug condition will administer cognitive assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metabolic Arm (Experimental): This arm includes a screening visit 1 and screening visit 2 to assess eligibility.
  This arm then includes the pancreatic euglycemic clamp procedure at visits 1 to 3. Visits 1 to 3 each consist of 3 days (day 0, day 1, and day 2).
  Olanzapine 2.5mg (or placebo) will be administered in doses of 5mg on day 0, 7.5mg on day 1, and 10mg on day 2.
  Day 2 consists of the final dose of olanzapine (or placebo) and the pancreatic euglycemic clamp procedure and other assessment procedures.
  On day 2, the participant is also randomized to and administered either intranasal insulin/Insulin Lispro 100 UNT/ML (or saline placebo) during the pancreatic euglycemic clamp procedure.
  Interventions: Drug: OLANZapine 2.5 MG; Drug: Placebo; Drug: Insulin Lispro 100 UNT/ML; Other: Saline
- Cognitive and MRI Arm (Experimental): This arm includes a screening visit 1 and screening visit 2 to assess eligibility. This arm includes an MRI scan and cognitive testing at visits 1 to 4. Visits 1 to 4 each consist of 3 days (day 0, day 1, and day 2).
  Olanzapine 2.5mg (or placebo) will be administered in doses of 5mg on day 0, and 10mg on day 1. Cognitive testing and MRI scanning then occur on day 2. On day 2, the participant is also randomized to and administered either intranasal insulin/Insulin Lispro 100 UNT/ML (or saline placebo) prior to conducting the MRI imaging and cognitive testing.
  Interventions: Drug: OLANZapine 2.5 MG; Drug: Placebo; Drug: Insulin Lispro 100 UNT/ML; Other: Saline

INTERVENTIONS:
Drug: OLANZapine 2.5 MG — Olanzapine capsules (2.5mg) will be administered with the following dosing schedules for each arm:
  1. Metabolic arm - 5mg on Day 0, 7.5mg on Day 1, and 10mg on Day 2
  2. Cognitive arm - 5mg on Day 0, 10mg on Day 1
  Other Names: Mylan-Olanzapine
Drug: Placebo — Placebo capsules visually identical to those containing olanzapine will be administered according to the same dosing schedule for each arm.
  Other Names: Olanzapine Placebo
Drug: Insulin Lispro 100 UNT/ML — Intranasal insulin spray (or placebo) will be administered on day 2 for each arm.
  For the metabolic arm: 40 IU of intranasal insulin lispro will be administered at timepoint 0 during the pancreatic euglycemic clamp procedure.
  For the cognitive arm: 160 IU of intranasal insulin lispro will be administered at about 11 am on day 2 prior to the MRI imaging and cognitive testing procedures.
  Other Names: Intranasal Insulin
Other: Saline — Placebo saline spray visually identical to the intranasal insulin spray will be administered on day 2 for each arm according the same dosing schedules.

SUMMARY:
Antipsychotic (AP) medications are considered to be the gold standard treatment for psychotic disorders including schizophrenia. However, APs have also been commonly associated with serious metabolic adverse effects including weight gain and Type 2 Diabetes, with younger populations disproportionately affected. In addition, young individuals treated with these agents have also been found to be at high risk for glucose dysregulation, including higher rates of prediabetes, with significant associations found between AP use and insulin resistance. Due to the concerning prevalence of these AP metabolic effects, it becomes important to further elucidate the mechanisms underlying AP effects on glucose metabolism, which are still poorly understood. One potential underlying mechanism is insulin which has been found to regulate hepatic (liver) glucose production through insulin receptors in the brain. These insulin receptors also play a role in neuronal growth and memory, or more broadly, cognition. Preliminary data in rat models has demonstrated that the AP olanzapine (OLA) inhibits the ability of a central insulin stimulus (acting at the level of the brain) to decrease endogenous glucose production (EGP), making this mechanism a prime target to translate from rodent models to human research. Furthermore, intranasal insulin (INI) administration (an analogous central insulin stimulus) has been repeatedly associated with improved cognitive performance for verbal memory and visuospatial functions in humans. Given these findings and with the goal of translational research, the present study will investigate OLA's effects in healthy human volunteers including: (a) the ability of INI to reduce EGP during a pancreatic euglycemic clamp (PEC; a glucose metabolism and insulin procedure); and (b) the ability of INI to improve cognitive performance. More specifically, the present study hypothesizes that:

1. INI will be associated with a decrease in EGP relative to intranasal placebo (INP) as measured by the PEC. This effect will be inhibited if OLA is co-administered.
2. OLA administration will be associated with decrements in cognitive measures (i.e., visuospatial, and verbal memory) as compared to placebo (PL). Additionally, OLA co-administration will block the beneficial effects of INI on cognition previously supported by other studies.
3. INI will result in adaptive changes in neurochemical and neurohemodynamic measures as studied using MRI imaging techniques.

DETAILED DESCRIPTION:
The primary objective of the study is to examine whether a single dose of OLA given to young healthy volunteers during PECs can inhibit the activity of a central insulin stimulus (i.e, INI) to reduce endogenous glucose production. Secondarily, in an exploratory arm, this study seeks to examine whether a single dose of OLA can inhibit improvements associated with INI administration on specific cognitive domains (visuospatial, and verbal memory). Further, the study will also explore the effects of insulin and OLA on neurochemical and neurohemodynamic measures obtained through MRI imaging techniques.

To accomplish these objectives, this study will have two separate and parallel arms - a metabolic PEC arm to study the primary hypothesis, and an MRI imaging and cognitive testing arm to study the two secondary hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-obese volunteers
* Age: 17 to 45 (Cognitive Arm) OR Ages 17-65 (Metabolic Arm)

Exclusion Criteria:

* History of current or past psychiatric illness (according to the Mini International Neuropsychiatric Interview [MINI]).[As an exception for the Metabolic Arm only, anxiety disorders will not be exclusionary (including, but not limited to: agoraphobia, social anxiety disorder, generalized anxiety disorder, and panic disorder)].
* Left-handedness (only for the cognitive and MRI arm)
* Pre-diabetes or diabetes (fasting glucose ≥6.0mmol/L or use of anti-diabetic drug);
* Evidence of impaired glucose tolerance on screening OGTT
* Family history of diabetes
* Use of weight reducing agents or other medications based on the discretion of the PI
* History of liver disease or AST> 2 times upper limit of normal
* History of kidney disease
* Major medical or surgical event within the last 6 months
* Any condition that interferes with safe acquisition of MRI data such as metal implants, pacemakers, cochlear implants, claustrophobia, etc. (only for the cognitive and MRI component)
* Pregnancy and/or breastfeeding

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Endogenous Glucose Production: Pancreatic Euglycemic Clamp Experiments | Visits 1-3 (12-16 weeks) for the metabolic arm
  Participants in the metabolic arm will complete four pancreatic euglycemic clamp (PEC) procedures. The PEC will measure changes in the ability of INI to reduce endogenous glucose production (EGP; the primary outcome measure) relative to INP and the presence of OLA (or PL). EGP will be reflected in dextrose infusion rates (InFR) measured during the PEC across treatment conditions.

SECONDARY OUTCOMES:
Changes in Cognitive Functioning: MRI scans across the 4 visit conditions | Visits 1-4 (9-18 weeks) for the cognitive arm
  Participants in the cognitive arm will complete 4 MRI scans that will include intra-scanner testing to assess changes in cognitive functioning across randomization conditions.
Oral Glucose Tolerance Test | Screening Visit 2 (1-2 weeks) for both arms
  Following collection of baseline samples, a standard glucose drink (75mg) is given orally, and a blood sample of insulin and glucose is obtained 2 hours after the glucose drink is administered. Serums which will be collected during this procedure include fasting glucose and fasting insulin related to weight gain and glucose metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Hahn, PhD, MD, Principal Investigator — Centre for Addiction and Mental Health; Satya Dash, MD, PhD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (2):
- Canada (2):
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Center for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stogios N, Hamel L, Smith E, Sanches M, Remington G, Voineskos A, Dash S, Graff-Guerrero A, Hahn M, Agarwal SM. Investigating the effects of antipsychotics on brain insulin action: Study protocol for a multi-modality magnetic resonance imaging (MRI) study in healthy controls. PLoS One. 2022 Nov 28;17(11):e0277211. doi: 10.1371/journal.pone.0277211. eCollection 2022. PMID 36441736